CLINICAL TRIAL: NCT01831479
Title: Investigation of Pharmacokinetic Interaction Between Rosuvastatin and Olmesartan in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Kyungsoo Park, Associate Professor, Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DWJ1276001
Record Dates: First submitted 2013-03-24; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics, drug-drug interaction
MeSH Terms: interventions — Rosuvastatin Calcium; olmesartan

ARMS (1):
- Rosuvastatin and Olmesartan (Experimental): A multiple-dose administration of rosuvastatin, a multiple-dose administration of olmesartan, and a multiple-dose administration of rosuvastatin and olmesartan, given orally with a washout period of 8 days between each administrations
  Interventions: Drug: Rosuvastatin; Drug: Olmesartan; Drug: Rosuvastatin and olmesartan

INTERVENTIONS:
Drug: Rosuvastatin — Single administration of rosuvastatin 20mg tablet QD for 7 consecutive days
Drug: Olmesartan — Single administration of olmesartan 40mg tablet QD for 7 consecutive days
Drug: Rosuvastatin and olmesartan — Co-administration of rosuvastatin 20mg tablet and and olmesartan 40mg tablet QD for 7 consecutive days

SUMMARY:
This study investigates pharmacokinetics and drug-drug interaction between Rosuvastatin and Olmesartan in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between the ages of 20 and 50 and within 20% of their ideal body weight, without congenital abnormality or chronic disease

Exclusion Criteria:

* History of cardiovascular, pulmonary, renal, endogenous, gastrointestinal, hematologic, neurologic or hemorrhagic disease;
* Clinically significant findings on routine laboratory (hematology, serum chemistry and urinalysis) or ECG tests;
* Use of prescription drugs in the 14 days immediately prior to starting the study that had the potential to interact with the study medication;
* Use of any substance that could induce or inhibit drug metabolism enzymes

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Profile of Pharmacokinetics | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72 hours post-dose with a sample at 72 hr being taken for rosuvastatin only
  Css,max, AUCtau

SECONDARY OUTCOMES:
Profile of Pharmacokinetics | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72 hours post-dose with a sample at 72 hr being taken for rosuvastatin only
  AUCss,last, AUCss,inf, Css,min, T_1/2

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea